CLINICAL TRIAL: NCT01383499
Title: A Phase II Randomised, Double-blind, Placebo-controlled Incomplete Crossover Trial With 4-week Treatment Periods to Evaluate Efficacy and Safety of Tiotropium Inhalation Solution (Doses of 1.25 µg, 2.5 µg and 5 µg) Delivered Via Respimat® Inhaler Once Daily in the Evening in Children 6 to 11 Yrs Old With Moderate Persistent Asthma
Brief Title: A Study to Evaluate Efficacy and Safety of Tiotropium in Children 6 to 11 Years Old With Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205.425; 2010-022458-18 (EudraCT Number)
Record Dates: First submitted 2011-06-20; First posted 2011-06-28 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Treatment A (Experimental): patients inhale 2 puffs (low dose) once daily in the evening via Respimat inhaler
  Interventions: Drug: Tiotropium bromide
- Treatment B (Experimental): patients inhale 2 puffs (medium dose) once daily in the evening via Respimat inhaler
  Interventions: Drug: Tiotropium bromide
- Treatment C (Experimental): patients inhale 2 puffs (high dose) once daily in the evening via Respimat inhaler
  Interventions: Drug: Tiotropium bromide
- Treatment D (Placebo Comparator): patients inhale 2 puffs of placebo inhalation solution matching tiotropium once daily in the evening via Respimat inhaler
  Interventions: Drug: Tiotropium bromide

INTERVENTIONS:
Drug: Tiotropium bromide — inhalation solution administered via Respimat in 3 different doses
  Arms: Treatment D
Drug: Tiotropium bromide — inhalation solution administered via Respimat in 3 different doses
  Arms: Treatment C
Drug: Tiotropium bromide — inhalation solution administered via Respimat in 3 different doses
  Arms: Treatment B
Drug: Tiotropium bromide — inhalation solution administered via Respimat in 3 different doses
  Arms: Treatment A

SUMMARY:
The aim of this trial is to select an optimum dose may be selected based on bronchodilator efficacy, safety evaluations and pharmacokinetics of tiotropium bromide.

ELIGIBILITY:
Inclusion criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment into this study:

1. All patients' parents (or legally accepted caregivers) must sign and date an informed consent prior to any study procedures including medication washout and restrictions. In addition, an informed assent suitable for this age group has to be obtained from patients.
2. Male or female patients between 6 and 11 years of age (up to 1 day prior to their 12th birthday at Visit 1).
3. All patients must have at least a 6-month history of asthma at the time of enrolment into the trial.
4. All patients must have been on maintenance treatment with inhaled corticosteroids at a stable medium dose - a patient is eligible on =200 µg to =400 µg Budesonide DPI or equivalent.
5. All patients must be symptomatic (partly controlled) at Visit 1 (screening) and prior to randomisation at Visit 2 as defined by an ACQ mean score of =1.5.
6. All patients must have a pre-bronchodilator FEV1 =60% and =90% of predicted normal at Visit 1. Variation of absolute FEV1 values of Visit 2 (pre-dose) as compared to values at Visit 2 (pre-bronchodilator) must be within ± 30%.
7. All patients must demonstrate an increase in FEV1 of =12% 15 to 30 min. after 200 µg salbutamol (albuterol) at Visit 1.
8. Patients must be able to inhale from the Respimat® inhaler correctly.
9. Patients must be able to perform all trial related procedures including technically acceptable spirometric manoeuvres according to current ATS/ERS standards and the use of the electronic diary/peak flow meter.

Exclusion criteria:

Patients with any of the following characteristics will not be eligible for entry into this study:

1. Patients with a significant disease other than asthma.
2. Patients with clinically relevant abnormal screening haematology or blood chemistry will be excluded if the abnormality defines a significant disease as defined in exclusion criterion 1. For participation in PK sampling, a haemoglobin of less than 11.3 g/dL will be regarded as exclusion criterion.
3. Patients with a history of congenital or acquired heart disease, or patients who have been hospitalised for cardiac syncope or failure during the past year.
4. Patients with any unstable or life-threatening cardiac arrhythmia, including cardiac arrhythmia requiring intervention (e.g. pacemaker implantation, catheter ablation etc.) or a change in drug therapy within the past year.
5. Patients with a malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years.
6. Patients with clinically significant lung diseases other than asthma, such as CF, or bronchopulmonary dysplasia.
7. Patients with known active tuberculosis.
8. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1.
9. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the 6 weeks prior to the screening visit (Visit 1).
10. Patients with known hypersensitivity to anticholinergic drugs, BAC, EDTA or any other components of the tiotropium inhalation solution.
11. Patients with known narrow-angle glaucoma, or any other disease where anticholinergic treatment is contraindicated.
12. Patients with moderate to severe renal impairment, as defined by a creatinine clearance <50 mL/min./1.73 m2 BSA, as tiotropium is a predominantly renally excreted drug.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (24):
- Germany (3):
  - 205.425.49005 Boehringer Ingelheim Investigational Site, Bochum
  - 205.425.49004 Boehringer Ingelheim Investigational Site, Dresden
  - 205.425.49002 Boehringer Ingelheim Investigational Site, Koblenz
- Hungary (4):
  - 205.425.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 205.425.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 205.425.36002 Boehringer Ingelheim Investigational Site, Mosdós
  - 205.425.36004 Boehringer Ingelheim Investigational Site, Szeged
- Latvia (6):
  - 205.425.37101 Boehringer Ingelheim Investigational Site, Baldone
  - 205.425.37105 Boehringer Ingelheim Investigational Site, Balvi
  - 205.425.37104 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.425.37106 Boehringer Ingelheim Investigational Site, Dubulti
  - 205.425.37102 Boehringer Ingelheim Investigational Site, Riga
  - 205.425.37103 Boehringer Ingelheim Investigational Site, Riga
- Lithuania (4):
  - 205.425.37004 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.425.37003 Boehringer Ingelheim Investigational Site, Tauragė
  - 205.425.37001 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.425.37002 Boehringer Ingelheim Investigational Site, Vilnius
- Russia (4):
  - 205.425.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 205.425.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 205.425.07001 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.425.07002 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Ukraine (3):
  - 205.425.38002 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.425.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 205.425.38003 Boehringer Ingelheim Investigational Site, Zaporizhya

REFERENCES:
- [Derived] Vogelberg C, Moroni-Zentgraf P, Leonaviciute-Klimantaviciene M, Sigmund R, Hamelmann E, Engel M, Szefler S. A randomised dose-ranging study of tiotropium Respimat(R) in children with symptomatic asthma despite inhaled corticosteroids. Respir Res. 2015 Feb 7;16(1):20. doi: 10.1186/s12931-015-0175-9. PMID 25851298

RESULTS

PARTICIPANT FLOW:
Groups:
- Tio R5/Placebo/Tio R1.25: Patients treated with Tiotropium 5 mcg in Period 1, with Placebo in Period 2 and with Tiotropium 1.25 mcg in Period 3. All products were administered once daily (QD) in the evening, delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication. No washouts (off treatment periods) between treatments.
- Tio R1.25/Tio R5/Tio R2.5: Patients treated with Tiotropium 1.25 mcg in Period 1, with Tiotropium 5 mcg in Period 2 and with Tiotropium 2.5 mcg in Period 3. All products were administered once daily (QD) in the evening, delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication. No washouts (off treatment periods) between treatments.
- Placebo/Tio R2.5/Tio R5: Patients treated with Placebo in Period 1, with Tiotropium 2.5 mcg in Period 2 and with Tiotropium 5 mcg in Period 3. All products were administered once daily (QD) in the evening, delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication. No washouts (off treatment periods) between treatments.
- Tio R2.5/Tio R1.25/Placebo: Patients treated with Tiotropium 2.5 mcg in Period 1, with Tiotropium 1.25 mcg in Period 2 and with Placebo in Period 3. All products were administered once daily (QD) in the evening, delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication. No washouts (off treatment periods) between treatments.
Period: Period 1 (4 Weeks)
Arm/Group | Tio R5/Placebo/Tio R1.25 | Tio R1.25/Tio R5/Tio R2.5 | Placebo/Tio R2.5/Tio R5 | Tio R2.5/Tio R1.25/Placebo
Started | 27 | 24 | 25 | 25
Completed | 26 | 24 | 25 | 25
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period 2 (4 Weeks)
Arm/Group | Tio R5/Placebo/Tio R1.25 | Tio R1.25/Tio R5/Tio R2.5 | Placebo/Tio R2.5/Tio R5 | Tio R2.5/Tio R1.25/Placebo
Started | 26 | 24 | 25 | 25
Completed | 26 | 24 | 25 | 25
Not Completed | 0 | 0 | 0 | 0
Period: Period 3 (4 Weeks)
Arm/Group | Tio R5/Placebo/Tio R1.25 | Tio R1.25/Tio R5/Tio R2.5 | Placebo/Tio R2.5/Tio R5 | Tio R2.5/Tio R1.25/Placebo
Started | 26 | 24 | 25 | 25
Completed | 26 | 24 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number of patients randomised and treated at all in the study.
Groups:
- Total.: Total number of patients randomised and treated at all in the study.
Arm/Group | Total.
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 69
Forced expiratory volume in 1s (FEV1) [Mean (Standard Deviation); unit: Litre] | 1.640 (0.386)

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume (FEV1) Peak (0-3h) Response
Description: The FEV1 peak (0-3h) response is determined at the end of the 4 week treatment period. This is the difference between the maximum FEV1 measured within the first 3 hours post dosing and the FEV1 baseline measurement. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: The Full analysis set (FAS) is defined as patients randomised, treated, with baseline data and at least one on-treatment efficacy measurement after 4 weeks on treatment within a period.
Measure: Least Squares Mean (Standard Error); unit: Litre
Groups:
- Placebo: Placebo once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
- Tio R1.25: Tiotropium 1.25 microgram once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
- Tio R2.5: Tiotropium 2.5 microgram once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
- Tio R5: Tiotropium 5 microgram once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 74 | 75
Litre | 0.185 (0.025) | 0.261 (0.026) | 0.290 (0.026) | 0.272 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Tio R5 minus Placebo; Test type: Superiority or Other; p = 0.0002, Mixed model repeated measures (MMRM) — First step of closed testing procedure, where the active treatments are compared to placebo. If this statistical test significant at the 0.05 alpha level then proceed to comparison of the next lower dose to placebo; This MMRM model includes treatment, period and baseline as fixed effects, and patient as random effect; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [0.042 to 0.132], Standard Error of Mean 0.023
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Tio R2.5 minus Placebo; Test type: Superiority or Other; p < .0001, Mixed model repeated measures (MMRM) — Second step of closed testing procedure. If this statistical test significant at the 0.05 alpha level then proceed to comparison of the next lower dose to placebo; This MMRM model includes treatment, period and baseline as fixed effects, and patient as random effect; Mean Difference (Final Values) = 0.104, 95% CI 2-sided [0.059 to 0.149], Standard Error of Mean 0.023
Statistical Analysis 3: Comparison: Placebo vs Tio R1.25; Tio R1.25 minus Placebo; Test type: Superiority or Other; p = 0.0011, Mixed model repeated measures (MMRM); This MMRM model includes treatment, period and baseline as fixed effects, and patient as a random effect; Mean Difference (Final Values) = 0.075, 95% CI 2-sided [0.030 to 0.120], Standard Error of Mean 0.023
Statistical Analysis 4: Comparison: Tio R1.25 vs Tio R5; Tio R5 minus Tio R1.25; Test type: Superiority or Other; Mixed model repeated measures (MMRM); Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.034 to 0.057], Standard Error of Mean 0.023
Statistical Analysis 5: Comparison: Tio R2.5 vs Tio R5; Tio R5 minus Tio R2.5; Test type: Superiority or Other; Mixed model repeated measures (MMRM); Mean Difference (Final Values) = -0.017, 95% CI 2-sided [-0.063 to 0.028], Standard Error of Mean 0.023
Statistical Analysis 6: Comparison: Tio R1.25 vs Tio R2.5; Tio R2.5 minus Tio R1.25; Test type: Superiority or Other; Mixed models repeated measures (MMRM); Mean Difference (Final Values) = 0.029, 95% CI 2-sided [-0.016 to 0.074], Standard Error of Mean 0.023

2. Secondary Outcome: Trough FEV1 Response
Description: The trough FEV1 is defined as the pre-dose FEV1 measured just prior to the last administration of randomised treatment. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with at least one on-treatment value.
Measure: Least Squares Mean (Standard Error); unit: Litre
Groups:
- Tio R1.25: Tiotropium 1.25 mcg once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
- Tio R2.5: Tiotropium 2.5 mcg once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
- Tio R5: Tiotropium 5 mcg once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 74 | 75
Litre | 0.085 (0.026) | 0.160 (0.026) | 0.190 (0.026) | 0.183 (0.026)

3. Secondary Outcome: Forced Vital Capacity (FVC) Peak (0-3h) Response
Description: The FVC peak (0-3h) response is determined at the end of the 4 week treatment period. This is the difference between the maximum FVC measured within the first 3 hours post dosing and the FVC baseline measurement. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with at least one on-treatment value.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 74 | 75
Litre | 0.202 (0.029) | 0.208 (0.029) | 0.253 (0.029) | 0.239 (0.029)

4. Secondary Outcome: FVC Trough Response
Description: The trough FVC response is defined as the pre-dose FVC measured just prior to the last administration of randomised treatment. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with at least one on-treatment value.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 74 | 75
Litre | 0.060 (0.030) | 0.109 (0.030) | 0.107 (0.030) | 0.113 (0.030)

5. Secondary Outcome: FEV1 Area Under the Curve From 0 to 3 h (AUC0-3h) Response
Description: FEV1 (AUC0-3h) will be calculated as the area under the curve from 0 to 3 hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with at least one on-treatment value.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 74 | 75
Litre | 0.110 (0.025) | 0.178 (0.025) | 0.208 (0.025) | 0.201 (0.025)

6. Secondary Outcome: FVC Area Under the Curve From 0 to 3 h (AUC0-3h) Response
Description: FVC (AUC0-3h) will be calculated as the area under the curve from 0 to 3 hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with at least one on-treatment value.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 74 | 75
Litre | 0.087 (0.027) | 0.097 (0.027) | 0.134 (0.027) | 0.110 (0.027)

7. Secondary Outcome: Mean Morning Peak Expiratory Flow (PEF) Response
Description: Mean morning PEF assessed by patients at home. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with at least one on-treatment value. For outcome measures obtained by AM3 device one patient in the "TioR2.5" group had no on-treatment data.
Measure: Least Squares Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 73 | 75
Litre/min | -0.928 (5.103) | 14.474 (5.127) | 12.045 (5.177) | 15.439 (5.127)

8. Secondary Outcome: Mean Evening PEF Response
Description: Mean Evening PEF assessed by patients at home. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 73 | 75
Litre/min | -0.568 (5.081) | 9.910 (5.103) | 6.991 (5.150) | 15.910 (5.103)

9. Secondary Outcome: Change From Baseline in the Number of Puffs of Rescue Medication Per Period (24 h, Daytime and Night-time Use)
Description: Mean number of inhalations (puffs) of unscheduled rescue salbutamol therapy during whole day (24 h, daytime and night-time use). Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 73 | 75
Puffs
  24 h | -0.664 (0.105) | -0.691 (0.105) | -0.314 (0.106) | -0.550 (0.105)
  Daytime | -0.338 (0.061) | -0.348 (0.062) | -0.130 (0.062) | -0.258 (0.062)
  Night-time | -0.354 (0.060) | -0.355 (0.060) | -0.180 (0.060) | -0.272 (0.060)

10. Secondary Outcome: Control of Asthma as Assessed by Asthma Control Questionnaire (ACQ)
Description: ACQ is a questionnaire consisting of seven point Likert scale ranging from 0 to 6, whereby 0 represents good control and 6 represents poor control of asthma. The scale describes the frequency and severity of asthma symptoms. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: 4 weeks
Population: FAS with at least one on-treatment value.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 74 | 75
Score | 0.966 (0.066) | 0.909 (0.066) | 0.846 (0.066) | 0.879 (0.066)

11. Secondary Outcome: Change From Baseline in Mean Number of Nighttime Awakenings
Description: Mean number of nighttime awakenings due to asthma symptoms as assessed by patients eDiary incorporated in the AM3® device. Analysis adjusted for treatment, period, patient and baseline using a mixed model. The scores for this question used the following scale where: 1='Did not wake up', 2='Woke up once', 3='Woke up 2-5 times', 4='Woke up more than 5 times' and 5='Was awake all night'.
Time Frame: Baseline and last week of treatment (week 4)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 76 | 75 | 73 | 75
scores on a scale | -0.135 (0.034) | -0.104 (0.034) | -0.080 (0.034) | -0.099 (0.034)

ADVERSE EVENTS:
Time Frame: 4 weeks + 30 days if in last period.
Description: All AEs, serious and non-serious, occurring during the course of the clinical trial were collected, documented, and reported to the sponsor by the investigator on the appropriate eCRF or SAE reporting forms.
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75 | 0/74 | 0/76
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75 | 0/74 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.